CLINICAL TRIAL: NCT04745338
Title: Effect Of Cryolipolysis On Visceral Adiposity Index In Polycystic Ovarian Syndrome Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Miral Saleh Mohamed, ASSISTANT LECTURER, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ECVAPP
Record Dates: First submitted 2021-02-03; First posted 2021-02-09 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- low caloric diet (Placebo Comparator): low caloric diet (1200cal/day)
  Interventions: Dietary Supplement: low calolric diet
- cryolipolysis (Active Comparator): cryolipolysis 3 sessions one session every 6 weeks by 3max cool shaping device
  Interventions: Device: 3max cool shaping device; Dietary Supplement: low calolric diet

INTERVENTIONS:
Device: 3max cool shaping device — cryolipolysis sessions are applied on abdomen area each session for 40 min. each
  Arms: cryolipolysis
Dietary Supplement: low calolric diet — low caloric diet (1200cal/day)

SUMMARY:
this study will be carried to investigate the effect of cryolipolysis on visceral adiposity index in pco women randomized controlled trial

DETAILED DESCRIPTION:
This study will be carried out on sixty females with polycystic ovarian syndrome (PCOS) who were selected from the Outpatient Clinic of Gynecology at Qasr Al Aini University Hospital. Their age ranged from 17-28 years, body mass index was 25-30 Kg/m2. They experienced hyperandrogenism, hyperinsulinemia and amenorrhea not less than 6 months.

PCOS females will be randomly assigned into two equal groups: group (A) (control group) consisted of 30 women who received low caloric diet (1200 Cal/day) and group (B) (study group) consisted of 30 women who received the same diet regime and cryolipolysis

ELIGIBILITY:
Inclusion Criteria:

* age ranges from 20-28 years, body mass index ranges 25-30 Kg/m2. They have pco syndrome .

Exclusion Criteria:

* Diabetic patients.
* Women with BMI>30
* Women having circulatory dysfunction.
* Women with respiratory or cardiac disease
* liver disease.
* Skin disease .
* Previous abdominal or uterine surgery
* Physical impairment

Ages: 20 Years to 28 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — it is carried on women with dysfunction in ovaries
Enrollment: 60 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2022-01-30 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Visceral adiposity index | 3 months
  indicator of adipose tissue distribution

SECONDARY OUTCOMES:
weight | up to 3 months
  anthropometric measurement by kilogram (kg)
waist circumference | up to 3 months
  anthropometric measurement by centimeter (cm)
high density lipoprotein | up to 3 months
  blood test
serum triglyceride level | up to 3months
  blood test

CONTACTS AND LOCATIONS:
Overall Officials: fahema me okiel, phd, Study Director — Cairo University; amal mo youssef, phd, Study Chair — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No